CLINICAL TRIAL: NCT03256318
Title: PLAY LONG: The Effect of Sports and Recreation Participation for Young chiLdren With physicAl disabilitY - Longitudinal Study
Brief Title: PLAY LONG: The Effect of Sports and Recreation Participation for Young chiLdren With physicAl disabilitY
Acronym: PLAY-LONG
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Nancy Flinn, Senior Scientific Advisor, Allina Health System
Other Study IDs: CKNF-1701
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Physical Disability; Quality of Life; Social Interaction; Health, Subjective

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children in Sports and Rec: Children with disabilities who enter the study between ages 5 and 10 who are participating in a Sports and Recreation Program. They will receive no intervention, only surveys.
  Interventions: Other: No intervention
- Comparison Children: Children with disabilities who enter the study between ages 5 and 10 and end participation in Sports and Recreation Program at a later date. They will receive no intervention, only surveys.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention; surveys/questionnaires only

SUMMARY:
Ten year longitudinal survey following children with disabilities who have participated in Sports and Recreation from a young age (5 to 10), and the parents of children who have participated in Sports and Recreation at a young age (5 to 10). These children will be followed for 10 years with surveys every 6 months, whether they are currently participating in sports and recreation activities or not.

The purpose of this longitudinal study is to examine the effects of early participation in organized sports and recreation activities (S&R) on self-reported health and health-related quality of life of children and youth (C&Y) with disabilities and their parent-reported social participation. This project will examine child and parent reported differences between:

1. C&Y with disabilities who participate in S&R and those who have discontinued participation in S&R programs
2. C&Y with disabilities who participate in sports vs. those who participate in recreation, and
3. C&Y with disabilities who participate in S&R and normative data on C&Y with disabilities and those without disabilities.

ELIGIBILITY:
Inclusion Criteria:

* At the time of enrollment, the child must be between the ages of 5 and 10 and be participating in an adapted sports and recreation program.
* At the time of enrollment, the parent must have a child between the ages of 5 and 10, who is participating in an adapted sports and recreation program.
* Children and parents who are enrolled in the study will continue to participate in the study for 10 years.

Exclusion Criteria:

* Children who are younger than 5 or older than 10 will not be entered into the study, nor will parents whose children are younger than 5 or older than 10 be entered into the study. .
* Individuals who do not read and write in English will be excluded from the study.
* Children who are wards of the state, or in foster care will be excluded from the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants for this research study will be recruited from five- to ten- year old children and their parents who are participating in adapted sports and recreation programs. These children will have a variety of physical disabilities, and be participating in a wide range of sports and recreation programs, including basketball, skiing, baseball, archery, bowling, curling, cycling, golf, horseback riding, martial arts, Nordic skiing, soccer, rock climbing, scuba, swimming, water skiing, rugby, softball tennis, and track and field. The types of sport and recreation activities changes from year to year, as activities become more or less popular.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Change in health related quality of life | Every 6 months for 10 years.
  As measured by KIDSCREEN-10 questionnaire

SECONDARY OUTCOMES:
Change in general health | Every 6 months for 10 years.
  Self reported general health as measured by PROMIS Pediatric Global Health Measure
Change in social participation | Every 6 months for 10 years.
  Self reported (or parent-reported) social participation as measured by PROMIS Pediatric Global Health Measure

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Flinn, PhD, OTR/L, Principal Investigator — Allina Health
Locations (1):
- Courage Kenny Rehabilitation Institute, Golden Valley, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No